CLINICAL TRIAL: NCT02754206
Title: Association Between Brain Blood Flow Regulation, Cognition, and Balance in Sports-Related Concussion
Brief Title: Cerebral Blood Flow Regulation and Concussions
Status: Terminated | Type: Observational
Why Stopped: PI left university and IRB protocol closed
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Heather McClary, Director of Research Compliance, Southern Methodist University
Other Study IDs: SouthernMethodist
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Brain Concussion; Post-Concussion Syndrome
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Subjects who are collegiate level athletes who do not have a concussion and are currently playing a contact-collision sport.
- Concussed: Subjects who have recently suffered a sports-related concussion and are currently a collegiate athlete playing a contact-collision sport.

SUMMARY:
The purpose of this study is to understand how biochemical markers in blood, balance disturbances, and cognitive performance are related to brain blood flow changes after a concussion.

DETAILED DESCRIPTION:
Comparisons will be made between control data and data following a concussion collected from athletes participating in contact-collision sports. For those suffering a concussion, comparisons will be made between day 3 (acute phase), day 21 (recovery phase), and 3 months post-concussion.

ELIGIBILITY:
Inclusion Criteria:

* Student athletes actively participating in collegiate sports. Subjects should be wiling to provide informed consent for participation in the study.

Exclusion Criteria:

* Participants who are unable to play as a result of injury. Presence of irregular heart beat.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Collegiate Athletes who are currently playing a contact-collision sport.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2016-01; Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow regulation | Change in Control, 3 days post concussion, 21 days post concussion, and 3 months post concussion
  Subject's cerebral blood flow regulation (cm/sec) at rest, during a cognitive test, and during a breathing test will be measured.

SECONDARY OUTCOMES:
Blood Biomarkers | Control, 3 days post concussion, 21 days post concussion, 3 months post concussion
  Subjects will have their blood drawn so investigators can look at biomarkers in their blood. The biomarkers will be Tau, a-Spectrin N-Terminal Fragment, Neuron-specific enolase, Ubiquitin C-Terminal hydrolase L1, S100B, and Glial fibrillary acidic protein.
Memory Function Test | Control, 3 days post concussion, 21 days post concussion, 3 months post concussion
  Subjects will be given paper tests to test their memory function.
Balance Test | Control, 3 days post concussion, 21 days post concussion, 3 months post concussion
  Subjects balance will be measured using a force plate.
Orthostatic Tolerance Test | Control, 3 days post concussion, 21 days post concussion, 3 months post concussion
  Subjects physiological measurements will be measured as the move from a seated position to a standing position.
Cerebral Vasoreactivity | Control, 3 days post concussion, 21 days post concussion, 3 months post concussion
  Subjects will breathe normal air, a 8% carbon dioxide gas mixture, and hyperventilate.

CONTACTS AND LOCATIONS:
Overall Officials: Sushmita Purkayastha, Ph.D, Principal Investigator — Southern Methodist University
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Purkayastha S, Adair H, Woodruff A, Ryan LJ, Williams B, James E, Bell KR. Balance Testing Following Concussion: Postural Sway versus Complexity Index. PM R. 2019 Nov;11(11):1184-1192. doi: 10.1002/pmrj.12129. Epub 2019 Apr 3. PMID 30729729